CLINICAL TRIAL: NCT01037283
Title: Feasibility of Interpersonal and Social Rhythm Therapy for Outpatients With Bipolar Disorder
Brief Title: Interpersonal and Social Rhythm Therapy Enter the Brief Title for Protocol IRB 09-003781>
Acronym: IPSRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Astrid Hoberg, Clinical Nurse Specialist, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-003781
Record Dates: First submitted 2009-12-18; First posted 2009-12-22 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Bipolar Disorder, Depressed
Keywords: Bipolar; Depressed
MeSH Terms: conditions — Bipolar Disorder; Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interpersonal and Social Rhythm Therapy (Other): All participants receive eight sessions of Interpersonal and Social Rhythm Therapy.
  Interventions: Behavioral: Interpersonal and Social Rhythm Therapy

INTERVENTIONS:
Behavioral: Interpersonal and Social Rhythm Therapy — Interpersonal and Social Rhythm Therapy delivered in two individual therapy sessions and six group therapy sessions.

SUMMARY:
In patients with bipolar disorder referred for psychotherapy, is interpersonal and social rhythm therapy delivered in a group psychotherapy format over 2-3 weeks feasible? This project will help determine if interpersonal social rhythm therapy can be delivered in the programmatic format being considered for the outpatient mood program.

ELIGIBILITY:
Adult patients with a confirmed diagnosis of Bipolar disorder in a depressed phase.

Referral for Interpersonal and Social Rhythm Therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Symptom improvement and patient satisfaction with group and programmatic format in the delivery of interpersonal and social rhythm therapy. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Hoberg, RN, CNS, Principal Investigator — Mayo Clinic